CLINICAL TRIAL: NCT02485002
Title: Differences in Urine Neutrophil Gelatinase-Associated Lipocalin (NGAL) Levels in Patients Undergoing Retrograde Intrarenal Surgery (RIRS) With or Without Ureteral Access Sheath (UAS)
Brief Title: Differences in Urine NGAL Levels in Patients Undergoing RIRS With or Without Ureteral Access Sheath
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Ozcan Kilic, Associate Professor, M.D., Selcuk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SU-RIRS-UAS-02
Record Dates: First submitted 2015-06-24; First posted 2015-06-30 (Estimated); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Urolithiasis
Keywords: kidney; kidney stone; NGAL; ureterorenoscopy; intrarenal surgery; kidney function
MeSH Terms: conditions — Urolithiasis; Kidney Calculi

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- UAS (+) (Active Comparator): RIRS with ureteral access sheath: A ureteral access sheath (UAS) will be positioned into the ureter of the patient prior to the insertion of the flexible ureterorenoscope (RIRS).
  Interventions: Device: RIRS with ureteral access sheath
- UAS (-) (Experimental): RIRS without ureteral access sheath: A ureteral access sheath (UAS) will not be positioned into the ureter of the patient prior to the insertion of the flexible ureterorenoscope (RIRS).
  Interventions: Device: RIRS without ureteral access sheath

INTERVENTIONS:
Device: RIRS with ureteral access sheath — Ureteral access sheath will be used during RIRS.
  Arms: UAS (+)
Device: RIRS without ureteral access sheath — Ureteral access sheath will not be used during RIRS.
  Arms: UAS (-)

SUMMARY:
This study will include patients aged between 18 and 65 who will undergo retrograde infrarenal surgery (RIRS) due to renal stone(s). A total of 60 patients (male or female) will be recruited, and will be randomized into 2 groups consisting of 30 patients in each group. The first group of patients will undergo RIRS with a ureteral access sheath (UAS) positioned prior to surgery; and the second group will undergo RIRS without UAS. As use of UAS decreases the pressure in the renal pelvis during RIRS, it is aimed to evaluate whether using UAS or not affects the kidney functions. besides the routine kidney function tests, namely urea and creatinine, neutrophil gelatinase-associated lipocalin (NGAL) (a more specific and early marker of kidney function) will be used to assess the differences in the kidney functions. Preoperative blood urea and creatinine levels and urine NGAL levels will be studied for all patients. After the surgery, blood urea and creatinine levels will be again studied as well as urine NGAL levels at postoperative 2nd hour, 72nd hour and 1st week.

ELIGIBILITY:
Inclusion Criteria:

* Being between 18-65 years old
* Having an indication of retrograde infrarenal surgery (RIRS) due to kidney stone

Exclusion Criteria:

* Patients with uncontrolled diabetes mellitus and diabetic nephropathy
* Patients with blood pressure > 140/80 mmHg despite regular use of antihypertensive agent(s)
* Patients with chronic kidney failure who need dialysis
* Patients who have had prerenal, renal or postrenal acute kidney failure 3 months or much earlier
* Patients who have had pyelonephritis 3 months or much earlier
* Patients younger than 18 years or older than 65 years
* Patients who have undergone a kidney surgery within the last 3 months and have abnormal kidney function tests
* Patients with a concomitant ureter stone who will undergo an endoscopic ureter stone treatment at the same session

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-06; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Urine NGAL level (ng/mL) | Within the first 7 days after surgery (RIRS)
  Determination of any impairment in renal function when ureteral access sheath is not used during RIRS by measuring urine NGAL level.

SECONDARY OUTCOMES:
Blood urea level (mg/dL) and creatinine level (mg/dL) | Within the first 7 days after surgery (RIRS)
  Determination of any impairment in renal function when ureteral access sheath is not used during RIRS by measuring blood urea and creatinine levels.

CONTACTS AND LOCATIONS:
Overall Officials: Ozcan Kilic, M.D., Principal Investigator — Selcuk University, School of Medicine, Department of Urology
Locations (1):
- Selcuk University, School of Medicine, Department of Urology, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Auge BK, Pietrow PK, Lallas CD, Raj GV, Santa-Cruz RW, Preminger GM. Ureteral access sheath provides protection against elevated renal pressures during routine flexible ureteroscopic stone manipulation. J Endourol. 2004 Feb;18(1):33-6. doi: 10.1089/089277904322836631. PMID 15006050
- [Background] Kourambas J, Byrne RR, Preminger GM. Does a ureteral access sheath facilitate ureteroscopy? J Urol. 2001 Mar;165(3):789-93. PMID 11176469
- [Background] L'esperance JO, Ekeruo WO, Scales CD Jr, Marguet CG, Springhart WP, Maloney ME, Albala DM, Preminger GM. Effect of ureteral access sheath on stone-free rates in patients undergoing ureteroscopic management of renal calculi. Urology. 2005 Aug;66(2):252-5. doi: 10.1016/j.urology.2005.03.019. PMID 16040093
- [Background] Stern JM, Yiee J, Park S. Safety and efficacy of ureteral access sheaths. J Endourol. 2007 Feb;21(2):119-23. doi: 10.1089/end.2007.9997. PMID 17338606
- [Background] Ichino M, Kusaka M, Kuroyanagi Y, Mori T, Morooka M, Sasaki H, Shiroki R, Shishido S, Kurahashi H, Hoshinaga K. Urinary neutrophil-gelatinase associated lipocalin is a potential noninvasive marker for renal scarring in patients with vesicoureteral reflux. J Urol. 2010 May;183(5):2001-7. doi: 10.1016/j.juro.2010.01.031. Epub 2010 Mar 19. PMID 20303517
- [Background] Abassi Z, Shalabi A, Sohotnik R, Nativ O, Awad H, Bishara B, Frajewicki V, Sukhotnik I, Abbasi A, Nativ O. Urinary NGAL and KIM-1: biomarkers for assessment of acute ischemic kidney injury following nephron sparing surgery. J Urol. 2013 Apr;189(4):1559-66. doi: 10.1016/j.juro.2012.10.029. Epub 2012 Oct 22. PMID 23085062